CLINICAL TRIAL: NCT01016106
Title: Genetic Screening for Filaggrin Mutation in Atopic Dermatitis and Ichthyosis Vulgaris in the African American Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: ViraCor Laboratories (Industry)
Responsible Party: Principal Investigator, Amy Paller, Professor and Chair of Department of Dermatology, Professor of Pediatrics, Northwestern University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: CMH 2010-14049
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Atopic Dermatitis; Ichthyosis Vulgaris
Keywords: eczema; atopic dermatitis; dry skin; ichthyosis vulgaris
MeSH Terms: conditions — Dermatitis, Atopic; Ichthyosis Vulgaris; Eczema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA pts AD and IV (Active Comparator): African American patients with a diagnosis of atopic dermatitis and ichthyosis vulgaris. During a single visit, a subject data collection form will be completed and DNA will be extracted from samples (buccal swabs) and then analyzed at IBT
  Interventions: Genetic: Buccal Swab
- AA patients (controls) (Active Comparator): African American patients with no personal or family history of ichthyosis vulgaris or atopy. During a single visit, a subject data collection form will be completed and DNA will be extracted from samples (buccal swabs) and then analyzed at IBT
  Interventions: Genetic: Buccal Swab

INTERVENTIONS:
Genetic: Buccal Swab — During a single visit, a subject data collection form will be completed and DNA will be extracted from samples (buccal swabs) and then analyzed at IBT laboratories in Lenexa, Kansas.

SUMMARY:
The investigators' primary objective is to identify common and rare mutations in the filaggrin gene in African American patients with a diagnosis of atopic dermatitis and ichthyosis vulgaris. Atopic dermatitis, or eczema, is a common, chronic, relapsing and remitting problem in many children and affects 10-20% of the pediatric population. Itch is a predominant feature of this disease and is quite disruptive to daily activities of life. In addition to itch, it is characterized by markedly dry skin, small red bumps that may have fluid. Ichthyosis vulgaris is characterized by extremely dry, scaly skin with a fine white scale and increased amounts of lines noted on the palms. Filaggrin is a protein that is essential for the skin to function properly as a barrier and found to be mutated in some European patients with ichthyosis vulgaris and atopic dermatitis. This association has not been looked at in the African American population. Genomic DNA (gDNA) will be purified from buccal swabs using commercially available kits and analyzed.

DETAILED DESCRIPTION:
Genetic screening and molecular dermatology allow physicians and scientists to screen populations who manifest a specific genetic disorder of skin, hair or nails and to study animal models for experiment-induced dermatopathology, diseases, and treatments. The purpose of such screening is to identify the gene(s) involved in eliciting the phenotypic characteristics that we as clinicians identify for diagnosis and treatment of said disease(s).

The field of genetics in dermatology has progressed immensely in the last 20 years and has strongly influenced the practice of dermatology. Most known single gene disorders, such as epidermoloysis bullosa, have been mapped to a particular chromosomal region and in many cases, the causative genes have been identified. However, more common diseases that are polygenic in origin such as atopic dermatitis remain a challenge to decipher. In addition, there still remain several monogenic disorders in which the underlying genetic basis is unclear.

In some cases, genetic analysis can be performed by sequencing entire genes or gene regions, or screening for specific common mutations. In the Japanese and some of the European populations, several researchers have been able to find an association between people with atopic dermatitis and ichythosis vulgaris and the filaggrin gene. Atopic dermatitis, or ezcema, is a common, chronic, relapsing and remitting problem in many children and affects 10-20% of the pediatric population. Atopic dermatitis is often called the itch that rashes, since itch is a predominant feature of this disease and is quite disruptive to daily activities of life. In addition to itch, it is characterized by markedly dry skin, small red bumps that may have fluid. Though treatments are available to help the rash resolve and to help with itch, this disease will continue to appear when treatments are stopped and often become infected.

Ichythosis vulgaris is quite prevalent, an estimated 1 in 250 persons are affected. It is characterized by extremely dry, scaly skin with a fine white scale and increased amounts of lines noted on the palms. Ichythosis vulgaris is thought to happen due to a combination of excess production of one of the layers of the skin and abnormal skin shedding.

Filaggrin is a protein that is essential for the skin to function properly as a barrier. It was initially thought to be one of the genes responsible for causing atopic dermatitis in 2006 after it was identified as the causal mutation in ichthyosis vulgaris. This association has been extensively studied in the European population and to a lesser extent in the Japanese population; however, has not been looked at in the African American population These new insights may help lead to future targeted therapy for these two extraordinarily common skin disorders.

General clinical applications of methods for diagnosis may include histological tissue examination, laboratory-based specimen analysis, and physical examination. However, although useful, all of these methods are limited to the identification of the phenotypic expression of the genetic abnormality. Conversely, genetic screening of tissue (collected via buccal swabs) enables the clinician and scientist to have access to a more finite method of diagnosis, treatment, and prevention options. Such methods of testing are particularly appealing for use in disorders in which the exact basis of the disease is unknown, as is the case of atopic dermatitis and ichythosis vulgaris in the African American population. Thus, genetic screening in the field of dermatology remains an important research agenda and is the focus of this proposal. This study allows for the collection of genetic material from patients seen in the dermatology clinic at Ann & Robert H Lurie Children's Hospital of Chicago.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 6 months
* Affected subjects: Must be African American and have a diagnosis of both atopic dermatitis or eczema as well as ichthyosis vulgaris
* Control subjects: Must be healthy African American subjects
* Must be willing to not apply emollients for 24 hours prior to visit.

Exclusion Criteria:

* Systemic illness
* Control subjects: Must not have a family history of atopy (including asthma, seasonal allergies or hay fever or allergic rhinitis, or eczema or atopic dermatitis)
* Control subjects: Must never have been given a diagnosis of eczema or atopic dermatitis
* Control subjects: Must not have excessively dry skin
* Must not be of Hispanic ethnicity

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2010-10 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Paller, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Ann & Robert H Lurie CHildren's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

REFERENCES:
- [Result] Polcari I, Becker L, Stein SL, Smith MS, Paller AS. Filaggrin gene mutations in African Americans with both ichthyosis vulgaris and atopic dermatitis. Pediatr Dermatol. 2014 Jul-Aug;31(4):489-92. doi: 10.1111/pde.12355. Epub 2014 Jun 12. PMID 24920311

RESULTS

PARTICIPANT FLOW:
Groups:
- African American (AA) Control Subjects: African American subjects with no personal or family history of ichthyosis vulgaris or atopy. Buccal swabs were obtained from each subject for deoxyribonucleic acid (DNA) analysis.
- AA Subjects With Atopic Dermatitis and Ichthyosis Vulgaris: African American subjects with a diagnosis of atopic dermatitis and ichthyosis vulgaris. Buccal swabs were obtained from each subject for deoxyribonucleic acid (DNA) analysis.
Period: Overall Study
Arm/Group | African American (AA) Control Subjects | AA Subjects With Atopic Dermatitis and Ichthyosis Vulgaris
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- African American (AA) Control Subjects: African American subjects with no personal or family history of ichthyosis vulgaris or atopy. Buccal swabs were obtained from each subject for DNA analysis.
- AA Subjects With Atopic Dermatitis and Ichthyosis Vulgaris: African American subjects with a diagnosis of atopic dermatitis and ichthyosis vulgaris. Buccal swabs were obtained from each subject for DNA analysis.
- Total: Total of all reporting groups
Arm/Group | African American (AA) Control Subjects | AA Subjects With Atopic Dermatitis and Ichthyosis Vulgaris | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 17 | 19
  Between 18 and 65 years | 8 | 1 | 9
  >=65 years | 7 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Heterozygous for Filaggrin (FLG) Null Mutations
Description: Buccal swab samples were obtained from each subject. Deoxyribonucleic acid (DNA) was purified from buccal swabs (IsoHelix Swabs, BocaScientific, Boca Raton, FL) and quantified by ultraviolet spectrophotometry. Purified genomic DNA and controls were amplified by polymerase chain reaction (PCR) from three different regions of FLG exon 3 with three primer sets. PCR products were analyzed by electrophoresis, purified (Qiaquick, Qiagen, Valencia, CA), and subjected to duplicate cycle sequencing reactions using ABI BigDye v3.1 reagents (Applied Biosystems, Carlsbad, CA). Labeled sequencing products were purified for capillary electrophoresis (ABI3730 or ABI3130 sequencer with POP7 polymer), and sequence results were examined using ABI SeqScape software. All nucleotide changes were noted, including 30 single nucleotide polymorphism (SNPs) in the population tested, the most common of which were coding changes at T454A, H2507Q, and G2545R, and silent change at nucleotide t2508c.
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | African American (AA) Control Subjects | AA Subjects With Atopic Dermatitis and Ichthyosis Vulgaris
Number analyzed (Participants) | 17 | 18
participants | 1 | 4

ADVERSE EVENTS:
Arm/Group | African American (AA) Control Subjects | AA Subjects With Atopic Dermatitis and Ichthyosis Vulgaris
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes